CLINICAL TRIAL: NCT00705042
Title: A Randomized, Open-Label, Single-Dose Administration, Parallel-Group, Multisite Study of the Pharmacokinetics of Etanercept, 25 or 50 mg, Administered Subcutaneously to Healthy Chinese Male Subjects
Brief Title: Study Evaluating Enbrel Drug Levels in Healthy Male Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0881A1-1110
Record Dates: First submitted 2008-06-17; First posted 2008-06-25 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 25 mg
  Interventions: Drug: Etanercept
- B (Experimental): 50 mg
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics (PK) and safety and tolerability of etanercept, 25 and 50 mg, administered as a single dose to healthy male Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy male Chinese subjects, ages 18 to 45. BMI in the range of 18 to 30 kg/m2 and weight greater than or equal to 50 kg.

Exclusion Criteria:

Active tuberculosis (TB) or history of TB. Serious infection (associated with hospitalization and/or antibiotics) within 1 month before study drug administration.

History of protein drug hypersensitivity.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
etanercept levels in the blood | 21 days

SECONDARY OUTCOMES:
Safety and tolerability of single doses of etanercept administered to healthy Chinese subjects | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- China (2):
  - Guangzhou, Guangdong
  - Beijing